CLINICAL TRIAL: NCT00544427
Title: Near Infrared Optical Coherence Tomography of the Upper Aero-Digestive Tract
Status: Withdrawn | Type: Observational
Why Stopped: Doesn't meet NIH clinical trial definition.
Sponsor: University of California, Irvine (Other)
Collaborators: Children's Hospital of Orange County (Other); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Brian Wong, M.D.,Ph.D Professor Department of Otolaryngology, University of California, Irvine
Other Study IDs: 20033025
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Disorder of Upper Digestive Tract
Keywords: Upper Areo-Digestive tract
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optical coherence tomography — Optical coherence tomography imaging

SUMMARY:
The Optical Coherence Tomography is a minimally-invasive diagnostic tool in both the office and operating room settings can identify sources of airway obstruction and effective surgical interventions. The researcher can use Optical Coherence Tomography to image tissues of the aero-digestive tract during surgical endoscopy in to the nose, oral cavity, larynx and ear in an outpatient clinic setting.

DETAILED DESCRIPTION:
The Optical Coherence Tomography imaging system has low power non-laser broad band infrared light shine onto laryngeal, esophageal, tracheal, oral, nasal and ear tissue and does not involve input of significant amounts of energy and no temperature rise occurs.

The gradual development and acceptance of Optical Coherence Tomography as an imaging modality serves as an alternative to invasive tissue biopsy as a diagnostic measure. Imaging diagnosis, can implement and more convenient than tissue biopsy and can reduce procedural complications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female age from new born to all age

Exclusion Criteria:

* subject who do not sign consent form

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be sekected from University of California Iriven Medical Cente department of Otolarygology/Head and neck surgery, Chao Digestive Diseases Center, Neonatal Intensive Care Unit and Beckman laser Institute and Children Hospital of Orange Pediatric Department.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic tool | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian JF Wong, M.D.,Ph.D., Principal Investigator — Beckman Laser Institute Medical Clinic,University ofCalifornia,Irvine
Locations (3):
- United States (3):
  - Beckman Laser Institute medical Clinic,University of California,Irvine, Irvine, California
  - Children Hospital of Orange, Orange, California
  - Otolaryngology-Head and Neck Surgery Medical Clinic,University of California,Irvine, Orange, California

REFERENCES:
- [Derived] Sharma GK, Ahuja GS, Wiedmann M, Osann KE, Su E, Heidari AE, Jing JC, Qu Y, Lazarow F, Wang A, Chou L, Uy CC, Dhar V, Cleary JP, Pham N, Huoh K, Chen Z, Wong BJ. Long-Range Optical Coherence Tomography of the Neonatal Upper Airway for Early Diagnosis of Intubation-related Subglottic Injury. Am J Respir Crit Care Med. 2015 Dec 15;192(12):1504-13. doi: 10.1164/rccm.201501-0053OC. PMID 26214043